CLINICAL TRIAL: NCT04266275
Title: An Investigation in the Use of Curcumin Topical Herbal Agent for the Treatment of Cervical Intraepithelial Neoplasia
Brief Title: Topical Curcumin for HPV Related Cervical Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lisa Flowers (Other)
Responsible Party: Sponsor-Investigator, Lisa Flowers, Professor, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00000758; IRB00117251 (Other: Emory Previous IRB number)
Record Dates: First submitted 2019-12-26; First posted 2020-02-12 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Neoplasm Cervix
Keywords: Cancer; HIV; Oncology; Infectious disease; HPV; Preventive medicine
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasms; Communicable Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Curcumin Arm (Experimental): Participants in this arm will use 2000 mg of intravaginal curcumin once a week for 20 weeks
  Interventions: Drug: Curcumin C3 Complex
- Placebo Arm (Placebo Comparator): Participants in this arm will use 2000 mg of intravaginal placebo once a week for 20 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Curcumin C3 Complex — Curcumin (Curcumin C3 Complex prepared by Sabinsa Corporation), a constituent of the spice turmeric, is considered to be a low-toxicity, dietary-derived agent with chemopreventative and therapeutic benefits.
  Study participants will be instructed to insert four 500 mg (2000 mg total) curcumin capsules once a week (excluding days when they are on their menses) for 20 weeks. Participants will insert capsules using the vaginal applicator while lying on their back with their knees bent. Participants will be instructed to gently insert the capsules into the vagina as far as they will go comfortably, similar to a tampon insertion or other common intravaginal drugs.
  Cervical cytology and HPV testing will be performed at baseline and 6 months after the baseline visit. If cervical cytology or HPV testing is abnormal at 6 months, a colposcopy with biopsies will be performed. All samples will be used to analyze for the study outcomes.
  Arms: Curcumin Arm
Drug: Placebo — Study participants randomized to the placebo arm will insert four 500 mg (2000 mg total) of the placebo (gelatin) capsules once a week (excluding days when they are on their menses) for 20 weeks. Participants will insert the capsules using the vaginal applicator while lying on their back with their knees bent. Participants will be instructed to gently insert the capsules into the vagina as far as they will go comfortably, similar to a tampon insertion or other common intravaginal drugs.
  Cervical cytology and HPV testing will be performed at baseline and 6 months after the baseline visit. If cervical cytology or HPV testing is abnormal at 6 months, a colposcopy with biopsies will be performed. All samples will be used to analyze for the study outcomes.
  Arms: Placebo Arm

SUMMARY:
The purpose of this study is to see if curcumin can suppress HPV infection in women with low-grade squamous intraepithelial lesions (LSIL) disease or treated high-grade squamous intraepithelial lesions (HSIL) disease. This study plans to explore the effect of curcumin as a potential medical treatment in HIV-uninfected and infected women with mild precancerous lesions of the cervix or recently treated high-grade precancerous lesions at risk for persistent HPV infection. About 200 women with low-grade precancerous lesions of the cervix or recently treated high-grade precancerous lesions will be enrolled to either insert 2000 mg of curcumin capsules in their vagina once a week or placebo after undergoing colposcopy or loop electrosurgical excision procedure (LEEP). They will have a repeat visit in 6 months where they will undergo a Pap smear and HPV test to determine if there are higher rates of HPV clearance after curcumin administration. If HPV is present or the Pap smear is abnormal, patients will then undergo colposcopic examination to evaluate cervical histology.

DETAILED DESCRIPTION:
Cervical cancer is the third most common cancer worldwide. The causative agent responsible for cervical cancer is the persistent infection with oncogenic Human Papillomavirus (HPV). Rates of cervical cancer and HPV infection are increased particularly in HIV-infected women due to immunosuppression with cervical cancer categorized as an AIDS-defining diagnosis. Despite the promise of HPV vaccine in the prevention of cervical cancer, the widespread availability of this vaccine is limited due to cost and accessibility. Therefore, prevention strategies to reduce the risk of cervical cancer after HPV exposure entail treatment at the premalignant state, including low-grade squamous intraepithelial lesions (LSIL) and high-grade squamous intraepithelial lesions (HSIL), along with the eradication of HPV infection. There is a desperate need for an inexpensive, non-invasive alternative method to treat these premalignant cervical lesions and potentially suppress HPV infection.

Curcumin, an extract from turmeric, a popular culinary spice, has been used in traditional Indian medicine for its anti-inflammatory and anti-infectious properties. Recent studies have shown the potential effect of curcumin to reduce tumors and precancerous lesions in animal and human cancer cells. It is postulated that curcumin achieves its effect on cancer cells by modulating different cellular pathways as well as altering HPV effect on tissue cells.

The purpose of this study is to see if curcumin can suppress HPV infection in women with LSIL disease or treated HSIL disease. The researchers plan to explore the effect of curcumin as a potential medical treatment in HIV-uninfected and infected women with mild precancerous lesions of the cervix or recently treated high-grade precancerous lesions at risk for persistent HPV infection. About 200 women with low-grade precancerous lesions of the cervix or recently treated high-grade precancerous lesions will be enrolled to either insert 2000 mg of curcumin capsules in their vagina once a week or placebo after undergoing colposcopy or LEEP. They will have a repeat visit in 6 months where they will undergo a Pap smear and HPV test to determine if there are higher rates of HPV clearance after curcumin administration. If HPV is present or the Pap smear is abnormal, patients will then undergo colposcopic examination to evaluate cervical histology.

ELIGIBILITY:
Inclusion Criteria:

* HIV-uninfected and infected women (without current AIDS-defining illness)
* Presence of a cervix
* Biopsy-proven LSIL disease or recently treated HSIL disease
* Adherence to combined anti-retrovirals (cART) if HIV infected
* On continuous antiretrovirals with a cluster of differentiation 4 (CD4) count >200 cells/ml with sustained undetectable viral load for at least 3 months (only for HIV-positive participants)
* On reliable birth control: combined oral contraceptive pills (OCP), long-acting reversible contraception (LARC), bilateral tubal ligation (BTL) or Depo-Provera (birth control shot)
* Willing to conform to the study requirements
* Reliable follow-up and contact information
* No risk factors for HSIL or microinvasive disease (no colposcopic features of microinvasion, adequate colposcopy and negative endocervical curettage)
* For women with HSIL only, LEEP completed within 6 weeks preceding initial encounter with study staff and adequate wound healing

Exclusion Criteria:

* Untreated HSIL or invasive features on colposcopy and the biopsy specimen
* Not adherent to anti-retroviral therapy (cART) (HIV infected participants)
* CD4 count =<200 cells/ml and detectable viral load within the last 3 months (only for HIV-positive participants)
* Lactating and pregnant people
* Patient with irregular cycles (more than once a month)
* Not on reliable birth control.
* Previous hysterectomy
* Prior diagnosis of cervical cancer, treated or untreated
* Inability to provide informed consent
* Medical condition that interferes with the conduct of the study in the investigator's opinion
* Evidence of active cervical infection or serious cervical disease necessitating surgery
* Known bleeding diathesis

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
HPV Clearance | Month 6
  HPV clearance, assessed as the number of participants with undetectable high-risk HPV mRNA levels in the standard monolayer Pap test (ThinPrep), at 6 months will be compared between the curcumin and placebo study arms.

SECONDARY OUTCOMES:
Disease Recurrence | Month 6
  Disease recurrence will be assessed either cytologic or histologic abnormality at 6 months. Rates of disease recurrence will be compared between study arms in HIV-uninfected and infected women.

OTHER OUTCOMES:
Participant Discontinuation | Month 6
  The treatment will be considered tolerable if 25% or fewer of participants discontinue the study early.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Flowers, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University, Atlanta, Georgia
  - Grady Memorial Hospital, Atlanta, Georgia
  - Grady Hospital - Ponce De Leon Clinic, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the published results will be made available for sharing after deidentification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available for sharing beginning 3 months and ending 5 years following article publication.
Access Criteria: Data will be available for sharing with researchers providing a methodologically sound proposal, in order to achieve aims in the approved proposal. Proposals should be directed to lflowe2@emory.edu. To gain access, data requestor will need to sign a data access agreement.